CLINICAL TRIAL: NCT03656965
Title: Randomized Phase III Study in EBV Positive Locally Advanced Nasopharyngeal Carcinoma Treated With Concurrent Chemo-radiotherapy With or Without Anti-Viral Drug
Brief Title: EBV Positive Nasopharyngeal Carcinoma Treated With Concurrent Chemo-radiotherapy With or Without Anti-Viral Drug
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Kuwait Cancer Control Center (Other)
Responsible Party: Principal Investigator, Khaled Alsaleh,MD, Chairman, Radiation Oncology Department, Kuwait Cancer Control Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RODKCCC
Record Dates: First submitted 2018-08-26; First posted 2018-09-04 (Actual); Last update posted 2018-09-04 (Actual); Status verified 2018-08

CONDITIONS: Drug Use for Unapproved Schedule
Keywords: EBV; Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Acyclovir; Radiotherapy; Drug Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Antiviral Drug with Chemoradiotherapy (Experimental): Antiviral therapy Acyclovir 800 mg per day during the whole course of treatment.
  Interventions: Drug: Acyclovir 800 MG; Combination Product: Radiotherapy and chemotherapy
- Chemoradiotherapy (Other): Patients will receive concurrent chemoradiotherapy which consisted of Cisplatin 40 mg/m2 weekly or 100mg/m2 every 3 weeks with IMRT 70Gy/35 fractions.
  Interventions: Combination Product: Radiotherapy and chemotherapy

INTERVENTIONS:
Drug: Acyclovir 800 MG — Acyclovir tablets 800 mg per day during the whole course of treatment Or Placebo.
  Arms: Antiviral Drug with Chemoradiotherapy
Combination Product: Radiotherapy and chemotherapy — Concurrent chemoradiotherapy which consisted of Cisplatin 40 mg/m2 weekly or 100mg/m2 every 3 weeks with IMRT 70Gy/35 fractions.

SUMMARY:
PCR-DNA of EBV test is a good prognostic indicator for survival after treatment (report: Prognostic Impact of Plasma, Epstein-Barr Virus DNA in Patients with Nasopharyngeal Carcinoma Treated using Intensity-Modulated Radiation Therapy.

The chances of the local recurrence or metastasis are higher in the patients at same stage with positive PCR-DNA of EBV in Nasopharyngeal carcinoma after same treatment.(ref.) Antiviral drugs have been used to inhibit EBV replication and target viral DNA polymerase are Foscarnet and phosphonoacetic acid both interact directly with the pyrophosphate-binding site of the enzyme, where Acyclovir as antiviral drug act at two levels: as competitive alternative substrates, competing with GTP on the substrate-binding site, and as DNA chain terminators, by incorporating into the growing DNA chain and blocking its elongation due to their acyclic structure.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed histopathologic diagnosis of nasopharyngeal squamous cell carcinoma, types WHO II-III.
* Stage II-IVB
* Requiring primary concomitant Radiotherapy and Chemotherapy.
* No head and neck surgery of the primary tumor or lymph nodes except for incisional or excisional biopsies.
* Positive PCR-DNA EBV
* ≥ 18 years of age
* ECOG performance status 0-1
* WBC ≥ 4,000/µl, platelets ≥ 100,000/µl; serum creatinine ≤ 1.6 mg/dl or 24 hr. calculated creatinine clearance ≥ 60 ml/min (see Section 3.1.6).
* Pre-treatment evaluation of tumor extent and tumor measurement.
* Nutritional and general physical condition must be considered compatible with the proposed radio-therapeutic treatment.
* Signed study-specific consent form prior to study entry Assessment.

Exclusion Criteria:

* Prior radiotherapy to the head and neck or any prior chemotherapy ≤ 6 months prior to study entry.
* Other malignancy except non-melanoma skin cancer or a carcinoma not of head and neck origin ≤ 5 years
* Evidence of distant metastasis.
* on any experimental therapeutic cancer treatment.
* major medical or psychiatric illness.
* pregnant females.
* Age ≤ 18 years old

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-05-01 (Actual); Primary Completion 2021-05 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Eliminated EBV titre as assessed by quantitative PCR-DNA in patients with NPC. | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Khaled AlSaleh, M.D, Principal Investigator — Chairman, Radiation Oncology Department
Locations (1):
- Kuwait Cancer Control Center, Kuwait City, Kuwait